CLINICAL TRIAL: NCT00271284
Title: A Crossover, Multicentre, Randomised Trial Comparing the Effect on the Control of Blood Glucose Concentration of Insulin Glargine and Insulin Detemir, Combined With Insulin Glulisine, Used as a Bolus, in Type 1 Diabetic Patients
Brief Title: Efficacy Study on the Control of Blood Glucose Concentration in Type 1 Diabetic Patients
Acronym: VARIABILITE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HMR1964A_3516; EudraCT #: 2005-002771-32
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin glulisine; Insulin Glargine; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental)
  Interventions: Drug: insulin glulisine / insulin glargine
- II (Active Comparator)
  Interventions: Drug: insulin glulisin / insulin detemir

INTERVENTIONS:
Drug: insulin glulisine / insulin glargine — insulin glargine administered subcutaneously by the patient once a day, in the evening, between 18.30 and 24.00
  Arms: I
Drug: insulin glulisin / insulin detemir — insulin detemir administered subcutaneously by the patient once a day, in the evening, between 18.30 and 24.00
  Arms: II

SUMMARY:
·Main objective: To compare the variability of fasting capillary blood glucose concentration, observed with insulin glargine combined with insulin glulisine and with insulin detemir combined with insulin glulisine, in type 1 diabetics. It is a non-inferiority study.

·Secondary objectives:

Efficacy:

* To compare the variability of blood glucose concentration before the evening meal, observed with insulin glargine combined with insulin glulisine and with insulin detemir combined with insulin glulisine, in type 1 diabetics.
* To record the intra- and inter-daily variability using the MAGE and MODD indices [1,2,3,4]
* To compare the glycaemic profiles (7 points)
* To evaluate the HbA1c concentration, at the end of each period of treatment, weight change, the dose of insulin used and the number of daily injections.

Tolerance:

* To record undesirable events
* To evaluate the safety in use from the record of episodes of hypoglycaemia (symptomatic, diurnal, nocturnal, severe).

ELIGIBILITY:
Inclusion Criteria :

* Belonging to a social security scheme or covered by such a scheme
* With type 1 diabetes (defined as a concentration of C-peptide < 0.1 nmol//l and a fasting blood glucose of >= 1.26 g/l), diagnosed not less than 5 years previously
* Treated for at least 6 months by intensive insulin treatment, following a basal-bolus system, using insulin glargine (Lantus®) as basal insulin. During the study, this insulin will administered in the evening
* Trained in the titration of prandial insulin (the dose of rapid insulin decided at each mealtime depending on the composition of the meal)
* With an HbA1c level of <= 8.5% at the inclusion visit
* Capable of checking their blood glucose concentration using the material supplied by the sponsor: blood glucose meter and patient notebook
* Able to eat 3 regular daily meals on the days for recording the blood glucose cycle and similarly as much as possible on other days throughout the length of the study
* Able to continue their usual daily activities during the study
* Women of child-bearing potential should be using an effective method of contraception
* Fundal examination result less than a year old available

Exclusion Criteria:

* Recent history of severe hypoglycaemia (at least 2 events in the 6 months prior to inclusion)
* An episode of acidocetosis in the 3 months prior to inclusion
* Proliferating retinopathy, defined as having required treatment by surgery or photocoagulation, in the 6 months prior to visit 1, or non-stabilised (rapidly developing) retinopathy which may require photocoagulation or surgery
* Pancreatectomy
* Altered hepatic function (AST or ALT >= 2.5 x normal, in the initial measurements)
* Altered renal function (plasma creatinine > 1.5 mg/dl)
* Acute infection
* Acute or chronic metabolic acidosis
* Gastroparesis
* History of cancer in the last 5 years
* Medically significant cardiovascular, hepatic, neurological or endocrine disease or any other significant disease making carrying out the protocol or interpreting the trial results difficult
* History of drug or alcohol abuse
* Subject likely to receive treatment during the trial which is not authorised in the protocol (see Section 6.2), in particular, treatment by corticosteroids whatever the route of administration or dose.
* Antidiabetic treatment by products other than those supplied within the framework of this study
* Treatment by another product undergoing development during the 3 months prior to inclusion in the trial
* Hypersensitivity to one of the study products (insulin glargine, insulin detemir, insulin glulisine) or to one of the excipients present in the insulin preparations, used in the study
* Working at night
* Pregnancy
* Breast-feeding
* Mental state making the subject incapable of understanding the objectives and possible consequences of the trial
* Subject unable to submit to the restrictions of the protocol (e.g. uncooperative, incapable of attending monitoring visits and probably incapable of finishing the trial)
* Subject deprived of his liberty because of an administrative or legal decision
* The investigator or any member of the team or close to the investigator directly implicated in the trial particularly assistant doctors, pharmacists, nurses, trial coordinator, etc.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2005-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Efficacy data : fasting blood glucose concentration | read daily during the last 2 months of each period

SECONDARY OUTCOMES:
Tolerance data : undesirable events including episodes of hypoglycaemia | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Marie SEBILLE, Dr, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Paris, France

REFERENCES:
- [Derived] Renard E, Dubois-Laforgue D, Guerci B; Variability Study Group. Non-inferiority of insulin glargine versus insulin detemir on blood glucose variability in type 1 diabetes patients: a multicenter, randomized, crossover study. Diabetes Technol Ther. 2011 Dec;13(12):1213-8. doi: 10.1089/dia.2011.0063. Epub 2011 Aug 2. PMID 21810024